CLINICAL TRIAL: NCT05871593
Title: CIRculating Cell-free nUcLeic Acids in Cancer Therapy Monitoring -01
Acronym: CIRCULATING-01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Consortium for Translational Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIRCULATING-01
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Next-Generation-Sequencing
Keywords: Next-Generation-Sequencing; Cell free DNA; Cell free RNA; Circulating tumor DNA; Circulating tumor RNA; Course of therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molecular genetic diagnostic (Other): Next-Generation-Sequencing (NGS)-methods
  Interventions: Genetic: Molecular genetic diagnostic

INTERVENTIONS:
Genetic: Molecular genetic diagnostic — With the help of modern, highly sensitive analysis methods (NGS), such as ultra-low high-throughput sequencing, even the smallest amounts of circulating cell-free nucleic acids in the blood can be detected. In the individual course of therapy, the changes in concentration of the tumor-specific variants can thus be continuously monitored and appropriate therapy decisions can be made. The presence of minimal residual diseases and the development of resistance mutations can also be examined using this technique.

SUMMARY:
In cooperation with the molecular tumor board of the University Hospital Tübingen (UKT), a prospective collection of blood samples during the course of therapy is planned. It is a pilot study in which the technical feasibility of the approach (Highly Sensitive Next-Generation Sequencing (NGS) methods) initially should to be evaluated and further developed.

DETAILED DESCRIPTION:
In this study, we would like to use and further develop Highly Sensitive Next-Generation Sequencing (NGS) methods. For this purpose, circulating cell-free nucleic acids (cell free desoxyribonucleic acid (cfDNA) or cell free ribonucleic acid (cfRNA)) are first isolated from the blood plasma. The circulating tumor desoxyribonucleic acid (ctDNA) and circulating tumor ribonucleic acid (ctRNA) fractions contained therein arise from the tumor tissue and can provide information about the existing tumor burden and the original tissue of the tumor. Somatic Single Nucleotide Variants (SNVs) and insertions and deletions (indels) serve as biomarkers within the ctDNA and ctRNA. The ctDNA also contains epigenetic information in the form of DNA methylation, which shows a characteristic pattern for each tissue. Informative regions of the genome can be specifically enriched using personalized or fixed NGS panels. In this way, an ultra-deep sequencing of defined regions can be carried out and even the smallest concentrations of ctDNA and ctRNA in liquid biopsies can be detected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Advanced tumor disease
* Ability to consent
* Existence of a declaration of consent signed by the patient and physician (informed consent for study participation and Comprehensive Cancer Center (CCC) biobank
* Existence or planned implementation of tumor-normal sequencing (usually carried out in a diagnostic context upon presentation at the Molecular Tumor Board (MTB)

Exclusion Criteria:

- No therapy recommendation by MTB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
cfDNA/cfRNA | Day 1: Preoperative
  Ratio of cfDNA/cfRNA preoperative
cfDNA/cfRNA | Day 2: At intervals of approx. 6-10 weeks
  Ratio of cfDNA/cfRNA during therapy
cfDNA/cfRNA | Day 3: Tumor recurrence or disease progression
  Ratio of cfDNA/cfRNA at recurrence or disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Schroeder, Dr., Principal Investigator — University Hospital Tübingen; Stephan Ossowski, Prof. Dr., Study Chair — University Hospital Tübingen

IPD SHARING:
Plan to Share IPD: Yes
The CIRCULATION-01 study will provide data in a pseudonymized manner to national and international databases set up to increase the diagnostic yield through advanced analysis tools.
Supporting Information: Analytic Code
Time Frame: Data will become available after analysis and unlimited.
Access Criteria: Authorized users within the participating organizations.